CLINICAL TRIAL: NCT03983850
Title: Phase I/II Study De-intensifying Exposure of Post-transplantation Cyclophosphamide as GVHD Prophylaxis After HLA-haploidentical Hematopoietic Cell Transplantation for Hematologic Malignancies
Brief Title: Optimizing PTCy Dose and Timing
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 190112; 19-C-0112
Record Dates: First submitted 2019-06-08; First posted 2019-06-12 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12-23

CONDITIONS: Graft Versus Host Disease; Hematologic Neoplasms
Keywords: Human Leukocyte Antigen; Busulfan; Fludarabine; Mycophenolate Mofetil; Sirolimus
MeSH Terms: conditions — Graft vs Host Disease; Hematologic Neoplasms | interventions — Busulfan; fludarabine; Cyclophosphamide; Mycophenolic Acid; Sirolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Donor Arm (No Intervention): Collection of bone marrow and/or PBSC (Up to 40 donors)
- Phase I Dose De-escalation (Experimental): PTCy at de-escalating doses (25 mg/kg/day on days +3 and +4, and PTCy 25 mg/kg on day +4) to assess for safety and determine Phase II dose (up to 12 evaluable patients)
  Interventions: Drug: Busulfan; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Mycophenolate Mofetil; Drug: Sirolimus
- Phase I duration de-escalation of MMF (Experimental): MMF at de-escalating duration (days +5 to +18 only, no MMF))
  Interventions: Drug: Busulfan; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Mycophenolate Mofetil; Drug: Sirolimus
- Phase I Pilot for Comparative Data (Experimental): Standard PTCy 50 mg/kg/day on days +3 and +4, in a small pilot (up to 5 evaluable patients) for comparative data
  Interventions: Drug: Busulfan; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Mycophenolate Mofetil; Drug: Sirolimus
- Phase II Efficacy (Experimental): PTCy at shortest duration, safe dose (from Phase I) to assess efficacy at providing adequate protection from grade 3-4 acute GVHD (up to 14 additional patients)
  Interventions: Drug: Busulfan; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Mycophenolate Mofetil; Drug: Sirolimus
- Phase II efficacy of reduced duration MMF (Experimental): MMF at duration identified from de-escalation evaluation.
  Interventions: Drug: Busulfan; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Mycophenolate Mofetil; Drug: Sirolimus

INTERVENTIONS:
Drug: Busulfan — Busulfan should be administered intravenously via a central venous catheter as a three-hour infusion every 24 hours.
  Arms: Phase I Dose De-escalation; Phase I Pilot for Comparative Data; Phase I duration de-escalation of MMF; Phase II Efficacy; Phase II efficacy of reduced duration MMF
Drug: Fludarabine — Fludarabine will be infused by IV over 60 minutes.
  Arms: Phase I Dose De-escalation; Phase I Pilot for Comparative Data; Phase I duration de-escalation of MMF; Phase II Efficacy; Phase II efficacy of reduced duration MMF
Drug: Cyclophosphamide — IV cyclophosphamide will be administered over 2 hours. Slower rates of infusion may be used to decrease side effects. A fluid intake of greater than 2 L/day is recommended during and for 1 to 2 days after cyclophosphamide administration.
  Arms: Phase I Dose De-escalation; Phase I Pilot for Comparative Data; Phase I duration de-escalation of MMF; Phase II Efficacy; Phase II efficacy of reduced duration MMF
Drug: Mycophenolate Mofetil — Any oral formulation should be taken on an empty stomach, 1 hour before or at least 2 hours after meals. Oral formulations should not be administered simultaneously with antacids. Avoid inhalation or direct contact with skin or mucous membranes of dry powder contained in capsules or suspension. IV solutions should be administered over at least two hours through either a peripheral or central vein and should not be administered by rapid or bolus injection.
  Arms: Phase I Dose De-escalation; Phase I Pilot for Comparative Data; Phase I duration de-escalation of MMF; Phase II Efficacy; Phase II efficacy of reduced duration MMF
Drug: Sirolimus — Oral tablets should be administered approximately 4 hours after cyclosporine administration. Sirolimus is administered orally, once daily, without food. Patients unable to tolerate tablets may take the oral solution formulation.
  Arms: Phase I Dose De-escalation; Phase I Pilot for Comparative Data; Phase I duration de-escalation of MMF; Phase II Efficacy; Phase II efficacy of reduced duration MMF

SUMMARY:
Background:

Stem cell or bone marrow transplants can cure or control blood cancers. Sometimes the donor cells see the recipient's body as foreign. This can cause complications. A high dose of the drug cyclophosphamide (PTCy) can help reduce these risks. Researchers want to see if a lower dose of PTCy can have the same benefits. Based on encouraging results from the first part of the study, researchers now are investigating whether a lower dose of PTCy can allow other immunosuppression to be decreased.

Objective:

To see if a lower dose of PTCy and now also shorter duration of another immunosuppressant called mycophenolate mofetil will help people with blood cancers have a more successful transplant and fewer side effects.

Eligibility:

People ages 15-65 with leukemia, lymphoma, or multiple myeloma that is not curable with standard therapy and is at high risk of returning without transplant, and their healthy adult relatives

Design:

Transplant participants will be screened with:

Blood, urine, breathing, and heart tests

Scans

Chest x-ray

Bone marrow samples: A needle inserted into the participant s pelvis will remove marrow and a bone fragment.

Transplant recipients will stay at the hospital and be prepped with chemotherapy over 6 days for the transplant. They will get stem cells through a catheter in the chest or neck. They will get the cyclophosphamide chemotherapy. They will stay in the hospital about 4 more weeks. They will have blood transfusions. They will have frequent blood tests and 2 bone marrow samples within 1 year after the transplant.

Donor participants will be screened with:

Blood, urine, and heart tests

Chest x-ray

Scans

Donor participants will have bone marrow taken from their pelvis or stem cells taken from their blood. For the blood donation, blood will be taken from a vein in one arm, move through a machine to remove white blood cells, and be returned through a vein in the other arm.

Participation will last up to 5 years....

DETAILED DESCRIPTION:
Background:

Post-transplantation cyclophosphamide (PTCy) reduces rates of severe acute and chronic graft-versus-host disease (GVHD) after allogeneic hematopoietic cell transplantation (HCT) and safely facilitates human leukocyte antigen (HLA)-haploidentical HCT

When clinically translated, the dose (50 mg/kg) and timing (days +3 and +4) of PTCy used were partly extrapolated from murine major histocompatibility complex (MHC)-matched skin allografting models and were partly empirical

In both MHC-haploidentical and MHC-disparate murine HCT models, a dose of 25 mg/kg/day was superior to 50 mg/kg/day on days +3 and +4 in terms of GVHD severity and mortality

In the MHC-haploidentical HCT model, a dose of 25 mg/kg on day +4 was equivalent to 25 mg/kg/day on days +3 and +4

In addition to better GVHD prevention, lower dosing of PTCy is associated with less broad reduction of T-cell numbers after PTCy

Mycophenolate mofetil (MMF), used as adjunct immunosuppression with standard dose PTCy, can have substantial gastrointestinal toxicity and can impede immune reconstitution and pathogen-specific immunity.

Objectives:

Determine whether a dose of PTCy 25 mg/kg on day +3 and +4 or on day +4 only can maintain adequate protection against grade III-IV acute GVHD.

Determine whether a reduced duration of MMF, in combination with PTCy 25 mg/kg/day on days +3 and +4, can maintain adequate protection against grade III-IV acute GVHD.

Eligibility:

Histologically or cytologically confirmed hematologic malignancy with standard indication for allogeneic hematopoietic cell transplantation including one of the following:

Acute myeloid leukemia (AML) of intermediate or adverse risk disease by the 2017 European LeukemiaNet criteria in first morphologic complete remission

AML of any risk in second or subsequent morphologic complete remission

B-cell acute lymphoblastic leukemia in first or subsequent complete remission

T-cell acute lymphoblastic leukemia with minimal residual disease detected after first line therapy and/or adverse genetics

Myelodysplastic syndrome of intermediate or higher score by the Revised International Prognostic Scoring System (IPSS-R)

Primary myelofibrosis of intermediate-2 or higher risk by the Dynamic International Prognostic Scoring System (DIPSS)

Chronic myelomonocytic leukemia

Chronic myelogenous leukemia resistant to or intolerant of >=3 tyrosine kinase inhibitors or with prior history of accelerated phase or blast crisis

B-cell lymphoma including Hodgkin lymphoma that has relapsed within 1 year of completion of primary treatment

Chronic lymphocytic leukemia with 17p deletion and/or unmutated IgHV or refractory to or intolerant of both BTK and PI3K inhibitors

Mature T or NK neoplasms as defined in the WHO guidelines of sufficient type and severity for allogeneic HCT based on the Prognostic Index for T-cell lymphoma (PIT) score of low-intermediate risk or higher or on recently published clinical practice guidelines

Hematologic malignancy of dendritic cell or histiocytic cell type

Multiple myeloma, stage III, relapsing after therapy with both a proteasome inhibitor and an immunomodulatory drug (IMiD)

Age 15-65.

At least one potentially suitable HLA-haploidentical donor.

Karnofsky performance score >=60

Adequate organ function

Design:

Open-label, single-center, non-randomized, phase I/II study

All patients will receive myeloablative conditioning, HLA-haploidentical bone marrow HCT, and GVHD prophylaxis with PTCy, MMF (depending on cohort), and sirolimus.

A small pilot of 5 evaluable patients will receive the standard PTCy 50 mg/kg on days +3/+4 to obtain a limited amount of comparative pharmacokinetic and T-cell immunophenotyping and repertoire data.

Then the study will proceed to a small, two-level [1) 25 mg/kg/day on days +3 and +4, 2) 25 mg/kg on day +4 only] phase I dose de-escalation study based on the standard 3+3 approach

Patients will be evaluated for development of grade III-IV acute GVHD (aGVHD) at day +60 as the dose-limiting toxicity and then phase II will proceed with the shorter duration of the days of treatment (+3/+4 or +4) which is associated with 0-1 of 6 patients with grade III-IV aGVHD at day +60 and with the least amount of toxicity

Simon optimal two-stage phase II trial design, to rule out excess grade III-IV acute GVHD with this decreased PTCy exposure, will be used in the phase II portion of the study which will enroll an additional 14 patients to see if this lower PTCy exposure is associated with a similar rate of grade III-IV acute GVHD as is expected with 50 mg/kg on days +3/+4

Following completion of the phase II portion of the trial evaluating PTCy 25 mg/kg/day on days +3/+4, a dose de-escalation will be conducted to determine if the dose of MMF (standardly days +5 to +35) may be reduced without meaningful impact on avoidance of grade III-IV acute GVHD. The tested dose levels will be 1) MMF from days +5 to +18 and 2) no MMF. This will be followed by a second Simon optimal two-stage phase II trial design, to rule out excess grade III-IV acute GVHD with decreased MMF exposure, which will expand on the lowest MMF dose that is associated with acceptable toxicity and enroll an additional 14 patients to see if this lower MMF is associated with a similar rate of grade III-IV acute GVHD as is expected with full 30 day MMF treatment.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion Criteria - Recipient

* Patients must have a histologically or cytologically confirmed hematologic malignancy with standard indication for allogeneic hematopoietic cell transplantation limited to one of the following:

  * Acute myeloid leukemia (AML) of intermediate or adverse risk disease by the 2017 European LeukemiaNet criteria in first morphologic complete remission (<5% blasts in the bone marrow, no detectable abnormal peripheral blasts, and no extramedullary disease)
  * AML of any risk in second or subsequent morphologic complete remission
  * B-cell acute lymphoblastic leukemia in first or subsequent complete remission
  * T-cell acute lymphoblastic leukemia with minimal residual disease detected after first line therapy and/or adverse genetics (no NOTCH1/FBXW7 mutation or presence of N/K-RAS mutation and/or PTEN gene alteration)
  * Myelodysplastic syndrome of intermediate or higher score by the Revised International Prognostic Scoring System (IPSS-R)
  * Primary myelofibrosis of intermediate-2 or higher risk by the DIPSS
  * Chronic myelomonocytic leukemia
  * Chronic myelogenous leukemia resistant to or intolerant of >=3 tyrosine kinase inhibitors or with history of accelerated phase or blast crisis
  * B-cell lymphoma including Hodgkin lymphoma that has relapsed within 1 year of completion of primary treatment
  * Chronic lymphocytic leukemia with 17p deletion and/or unmutated IgHV or refractory to or intolerant of both BTK and PI3K inhibitors
  * Mature T or NK neoplasms as defined in the WHO guidelines of sufficient type and severity for allogeneic HCT based on the Prognostic Index for T-cell lymphoma (PIT) score of low-intermediate risk or higher or on recently published clinical practice guidelines
  * Hematologic malignancy of dendritic cell or histiocytic cell type
  * Multiple myeloma, stage III, relapsing after therapy with both a proteasome inhibitor and an immunomodulatory drug (IMiD)
* Age 15-65. Patients <18 years old must be at least 50 kg. Note: Because patients 15-17 years old and <50 kg are not able to be cared for on the adult oncology wards and by the investigative team, they are excluded.
* At least one potentially suitable HLA-haploidentical donor.
* Karnofsky performance score >=60
* Adequate organ function defined as possessing all of the following:

  * Cardiac ejection fraction >=45% by 2D ECHO;
  * Forced expiratory volume-1 (FEV-1), forced vital capacity (FVC), and diffusing capacity of the lung for carbon monoxide (DLCO) (corrected for hemoglobin) all of >=50% predicted;
  * Estimated serum creatinine clearance of >=60 ml/minute/1.73m^2 calculated using eGRF in the clinical lab for adults and the Schwartz formula for pediatric subjects;
  * Total bilirubin <=2X the upper limit of normal;
  * Alanine aminotransferase and aspartate aminotransferase <=3X the upper limit of normal.
* Myeloablative conditioning is toxic to the developing human fetus and is teratogenic. For this reason, the following measures apply:

  * Individuals of child-bearing potential (IOCBP) and participants who can father children must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for at least one year post-transplant.
  * IOCBP must have a negative serum or urine pregnancy test within 7 days prior to enrollment.
* Ability of subject or Legally Authorized Representative to understand and the willingness to sign a written informed consent document. Pediatric patients (<18 years of age) will provide assent, and the parent(s) or legal guardian(s) will provide informed consent.
* Subjects requiring standard therapies to prepare for HCT should be referred in remission if possible. However, these diseases are often aggressive and require swift evaluation for HCT while concurrently attempting to establish disease control through the administration of standard therapies. If ongoing therapy for the underlying disease outside of the NIH is not in the best interest of the subject according to the clinical judgment of the PI, then the subject may receive up to 2 cycles of standard treatment for his/her underlying hematologic malignancy as a bridge to HCT on this protocol, prior to starting the research phase of the study. The subject must have a Karnofsky performance status of >= 60% at the start of the first cycle to proceed. If it becomes apparent that the subject will not be able to proceed to HCT, then he/she must come off study. Subjects receiving standard therapy will be told about the therapy, associated risks, potential benefits, alternatives to the proposed therapy, and the availability of receiving the same treatment elsewhere, outside of a research protocol.

EXCLUSION CRITERIA:

Exclusion Criteria - Recipient

* Patients who are receiving any other investigational agents. Prior experimental therapies must have been completed at least 4 weeks prior to the date of beginning conditioning.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection excluding controlled fungal infection on appropriate treatment, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, endocrinopathy (significant uncontrolled or untreated hypothyroidism, hyperthyroidism, or adrenal insufficiency), or active psychiatric illness/social situations that would limit compliance with study requirements
* Prior myeloablative conditioning for autologous or allogeneic HCT.
* An HLA-matched-sibling donor who is available and willing to donate bone marrow. Note: The patient must have access to HCT using this donor for this to be an exclusion criterion.
* Individuals who are pregnant or who intend to become pregnant during the study are excluded because myeloablative conditioning is toxic to the developing fetus with the potential for teratogenic or abortifacient effects.
* Nursing participants must be willing to discontinue nursing at the time of the study treatment initiation, as the potential for some of the study medications to be transmissible via nursing is unknown.
* Active malignancy of non-hematopoietic type (excluding non-melanoma skin cancers) which is: metastatic, or relapsed/refractory to treatment, or locally advanced and not amenable to curative treatment, or limited disease treated with curative intent treatment within the last 2 years. This excludes non-melanoma skin cancers.
* The severity of the hematologic malignancy does not warrant the potential toxicity of myeloablative allogeneic HCT as judged by the PI.

INCLUSION CRITERIA:

Inclusion Criteria - Related Donor

* Related donor deemed suitable and eligible, and willing to donate, per clinical evaluations, who are additionally willing to donate blood, bone marrow, saliva, oral swab, and stool for research. Related donors will be evaluated in accordance with existing institutional Standard Policies and Procedures for determination of eligibility and suitability for clinical donation.
* Ages >= 12 years

EXCLUSION CRITERIA:

Exclusion Criteria - Related Donor

-None

Ages: 12 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2026-10-26 (Estimated)

PRIMARY OUTCOMES:
aGVHD protection from a reduced duration of MMF, in combination with PTCy 25 mg/kg/day | 60 days
  The fraction of evaluable patients who experience grade III-IV aGVHD at day +60 will be determined and reported along with 80% and 95% two-sided confidence intervals. The MMF duration level patients may be compared with the PTCy dose level patients which serves as a baseline for standard duration MMF.
aGVHD protection from PTCy 25 mg/kg | 60 days
  The fraction of evaluable patients who experience grade III-IV aGVHD at day +60 will be determined and reported along with 80% and 95% two-sided confidence intervals.

SECONDARY OUTCOMES:
Determine, at the PTCy dose or MMF duration used in phase II cohorts, the cumulative incidences | 100 days
  Rate and timing of neutrophil and platelet engraftment also will be evaluated descriptively, including fractions who attain each condition at day 28 and 100, along with 95% confidence intervals. Ranges and medians will be calculated only in engrafting patients. Grade II-IV aGVHD also will be evaluated descriptively including fractions who attain each condition at day 100 and 200 days, and 95% confidence intervals. Grade III-IV aGVHD also will be evaluated descriptively including fractions who attain each condition at day 100 and 200 days, and 95% confidence intervals
determine the shortest MMF duration without unacceptable acute GVHD to be used during phase II | 60 days
  The phase II MMF duration level patients may be compared with the phase II PTCy dose level patients which serves as a baseline for standard duration MMF.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher G Kanakry, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared. @@@@@@@@@@@@All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Data from this study may be requested by contacting the PI.@@@@@@@@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Derived] Hyder MA, Dimitrova D, Sabina R, DeVries A, McCune JS, McAdams MJ, Flomerfelt FA, McKeown C, Sadler JL, Chai A, Hughes TE, Napier S, Stokes A, Sponaugle J, Rechache K, Parta M, Cuellar-Rodriguez J, Figg WD, Choo-Wosoba H, Steinberg SM, Kanakry JA, Kanakry CG. Intermediate-dose posttransplantation cyclophosphamide for myeloablative HLA-haploidentical bone marrow transplantation. Blood Adv. 2025 May 27;9(10):2553-2569. doi: 10.1182/bloodadvances.2024014879. PMID 39908565
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-C-0112.html